CLINICAL TRIAL: NCT04470908
Title: A Phase 1, Open-label, Fixed-sequence Study to Investigate the Effect of the Moderate CYP3A Inducer Rifabutin on the Pharmacokinetics of Zanubrutinib in Healthy Male Subjects
Brief Title: The Effect of Moderate CYP3A Inducer Rifabutin on the Pharmacokinetics of Zanubrutinib in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-112
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Male
Keywords: Phase 1; Healthy volunteers; Pharmacokinetics
MeSH Terms: interventions — zanubrutinib; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib + Rifabutin (Experimental): Day 1: zanubrutinib
  Days 3 to 10: rifabutin
  Day 11: zanubrutinib and rifabutin
  Interventions: Drug: Zanubrutinib; Drug: Rifabutin

INTERVENTIONS:
Drug: Zanubrutinib — Single oral dose of 320 mg
  Other Names: BGB-3111; Brukinsa
Drug: Rifabutin — Oral dose of 300 mg once daily

SUMMARY:
The primary objective of this study was to determine the effect of the moderate cytochrome P450 3A (CYP3A) inducer rifabutin on the pharmacokinetics (PK) of zanubrutinib in healthy males.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males of any race, between 18 and 65 years of age, inclusive.
2. Male participants in good health as determined by past medical history, physical examination, vital signs, ECG and laboratory tests at screening
3. Must have a body mass index (BMI) between 18 and 32 kg/m^2

Key Exclusion Criteria:

1. Participants with a clinically relevant history or presence of any clinically significant disease
2. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy, cholecystectomy, and hernia repair will be allowed)
3. History of drug or alcohol abuse within 1 year prior to check-in
4. Use or intended use of any nonprescription medications/products including vitamins, minerals, herbal/plant-derived preparations within 7 days prior to check-in
5. A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result and/or a positive human immunodeficiency virus (HIV) at screening
6. Use of tobacco- or nicotine-containing products within 3 months prior to check-in
7. Use or intended use of any prescription medications/products within 14 days prior to check-in

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tariq B, Conto S, Cohen A, Sahasranaman S, Ou YC. A Phase 1, Open-Label, Fixed-Sequence, Drug-Drug Interaction Study of Zanubrutinib with Rifabutin in Healthy Volunteers. Clin Pharmacol Drug Dev. 2023 Aug;12(8):832-838. doi: 10.1002/cpdd.1250. Epub 2023 May 5. PMID 37145975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center study with dosing in a fixed sequence. A total of 13 participants were enrolled and 12 completed the study.
Groups:
- Zanubrutinib + Rifabutin: Single oral dose zanubrutinib 320 mg on Days 1 and 11 in the fasted state and once daily oral rifabutin 300 mg on Days 3 to 10 with food and on Day 11 in the fasted state
Period: Zanubrutinib on Day 1
Arm/Group | Zanubrutinib + Rifabutin
Started | 13
Completed | 13
Not Completed | 0
Period: Rifabutin on Days 3 to 10
Arm/Group | Zanubrutinib + Rifabutin
Started | 13
Completed | 13
Not Completed | 0
Period: Zanubrutinib + Rifabutin on Day 11
Arm/Group | Zanubrutinib + Rifabutin
Started | 13
Completed | 12
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zanubrutinib + Rifabutin
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.8 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Zanubrutinib
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose on Days 1 and 11
Population: The pharmacokinetic (PK) population included all participants who received at least 1 dose of zanubrutinib and had evaluable PK data (at least 1 PK parameter could be calculated).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Zanubrutinib: Single oral dose zanubrutinib 320 mg on Day 1 (reference)
- Zanubrutinib + Rifabutin: Single oral dose zanubrutinib 320 mg on Day 1 and after co-administration with oral rifabutin 300 mg on Day 11 (test)
Arm/Group | Zanubrutinib | Zanubrutinib + Rifabutin
Number analyzed (Participants) | 13 | 13
h*ng/mL | 2700 (24.8) | 1530 (21.4)
Statistical Analysis 1: Comparison: Zanubrutinib vs Zanubrutinib + Rifabutin; Test type: Other — Estimate the geometric least square mean ratio of Zanubrutinib vs Zanubrutinib + Rifabutin; Ratio of Geometric Least Squares Means = 0.566, 90% CI 2-sided [0.525 to 0.610]

2. Primary Outcome: AUC From Time Zero to Infinity (AUC0-∞) of Zanubrutinib
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose on Days 1 and 11
Population: The PK population included all participants who received at least 1 dose of zanubrutinib and had evaluable PK data (at least 1 PK parameter could be calculated).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Zanubrutinib | Zanubrutinib + Rifabutin
Number analyzed (Participants) | 13 | 12
h*ng/mL | 2780 (23.3) | 1590 (22.2)
Statistical Analysis 1: Comparison: Zanubrutinib vs Zanubrutinib + Rifabutin; Test type: Other — Estimate the geometric least square mean ratio of Zanubrutinib vs Zanubrutinib + Rifabutin; Ratio of Geometric Least Squares Means = 0.560, 90% CI 2-sided [0.532 to 0.589]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Zanubrutinib
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose on Days 1 and 11
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Zanubrutinib | Zanubrutinib + Rifabutin
Number analyzed (Participants) | 13 | 13
ng/mL | 489 (38.1) | 253 (33.7)
Statistical Analysis 1: Comparison: Zanubrutinib vs Zanubrutinib + Rifabutin; Test type: Other — Estimate the geometric least square mean ratio of Zanubrutinib vs Zanubrutinib + Rifabutin; Ratio of Geometric Least Squares Means = 0.518, 90% CI 2-sided [0.441 to 0.608]

4. Primary Outcome: Time to the Maximum Observed Plasma Concentration (Tmax) of Zanubrutinib
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose on Days 1 and 11
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Zanubrutinib | Zanubrutinib + Rifabutin
Number analyzed (Participants) | 13 | 13
Hours | 1.50 [1.00 to 4.02] | 2.00 [1.00 to 8.00]

5. Primary Outcome: Time of the Last Quantifiable Concentration (Tlast) of Zanubrutinib
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose on Days 1 and 11
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Zanubrutinib | Zanubrutinib + Rifabutin
Number analyzed (Participants) | 13 | 13
Hours | 36.0 [24.0 to 36.0] | 36.0 [24.0 to 36.0]

6. Primary Outcome: Apparent Terminal Elimination Half-life (t1/2) of Zanubrutinib
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose on Days 1 and 11
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Zanubrutinib | Zanubrutinib + Rifabutin
Number analyzed (Participants) | 13 | 12
Hours | 7.24 (3.10) | 7.00 (4.46)

7. Primary Outcome: Apparent Oral Clearance (CL/F) of Zanubrutinib
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose on Days 1 and 11
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Zanubrutinib | Zanubrutinib + Rifabutin
Number analyzed (Participants) | 13 | 12
Liters/hour | 115 (23.3) | 201 (22.2)

8. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Zanubrutinib
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose on Days 1 and 11
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Zanubrutinib | Zanubrutinib + Rifabutin
Number analyzed (Participants) | 13 | 12
Liters | 1080 (68.4) | 1750 (70.9)

9. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: Adverse events (AEs) and serious adverse events included for summary, AEs that start during or after the first dose, or start prior to the first dose and increases in severity after the first dose, including vital signs, physical examination, electrocardiogram, and laboratory parameters
Time Frame: From the date of first study drug administration to 30 days after last dose (up to 3.5 months)
Population: The safety population included all participants who received at least 1 dose of zanubrutinib.
Measure: Count of Participants; unit: Participants
Groups:
- Zanubrutinib on Day 1: Single oral dose zanubrutinib 320 mg on Day 1
- Rifabutin on Days 3 to 10: Once daily oral rifabutin 300 mg on Days 3 to 10
- Zanubrutinib + Rifabutin on Day 11: Single oral dose zanubrutinib 320 mg and once daily oral rifabutin 300 mg on Day 11
Arm/Group | Zanubrutinib on Day 1 | Rifabutin on Days 3 to 10 | Zanubrutinib + Rifabutin on Day 11
Number analyzed (Participants) | 13 | 13 | 13
Participants
  At least 1 treatment-emergent adverse event (TEAE) | 1 | 6 | 0
  Serious adverse events | 0 | 0 | 0
  Vital sign TEAEs | 0 | 0 | 0
  Physical examination TEAEs | 0 | 0 | 0
  Electrocardiogram TEAEs | 0 | 0 | 0
  Laboratory-related TEAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of first study drug administration to 30 days after last dose (up to 3.5 months)
Description: The safety population included all subjects who received at least 1 dose of zanubrutinib
Arm/Group | Zanubrutinib on Day 1 | Rifabutin on Days 3 to 10 | Zanubrutinib + Rifabutin on Day 11
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 6/13 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zanubrutinib on Day 1 (N=13) | Rifabutin on Days 3 to 10 (N=13) | Zanubrutinib + Rifabutin on Day 11 (N=13)
Chromaturia (Renal and urinary disorders) | 0 (0) | 6 (6) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT04470908/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04470908/SAP_001.pdf